CLINICAL TRIAL: NCT01820650
Title: A Prospective, Multicenter Study to Evaluate the ConforMIS iTotal® (CR) Knee Replacement System
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-001
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee replacement; patient-specific
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: iTotal G2 CR Knee Replacement System — Total Knee replacement

SUMMARY:
This study is designed to observe the long term clinical outcomes of patient-specific knee arthroplasty in patients with osteoarthritis.

DETAILED DESCRIPTION:
If the patient has previously received a standard total knee replacement in their contralateral knee, the primary endpoint questionnaire and some secondary endpoint questionnaires will be completed regarding BOTH their iTotal® CR knee and their standard total knee for all time points where questionnaires are required by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition included in the approved Indications For Use for the iTotal® CR
* Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a TKR procedure. Disease status is assessed by Clinical and Radiographic assessment.
* Willingness to participate in the clinical study, to give informed consent and to attend all follow-up visits
* > 18 years of age

Exclusion Criteria:

* Simultaneous bilateral procedure required
* BMI > 40
* Active malignancy (defined as a history of any invasive malignancy - except non-melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
* Poorly Controlled diabetes
* Neuromuscular conditions which prevent patient from participating in study activities
* Active local or systemic infection
* Immunocompromised
* Fibromyalgia or other general body pain related condition
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated to an extent that the procedure is unjustified
* Diagnosed with or receiving treatment for Osteoporosis
* Other physical disability affecting the hips, spine, or contralateral knee.
* Severe instability due to advanced loss of osteochondral structure
* Prior arthroplasty of the affected knee, including High Tibial Osteotomy (HTO)
* Compromised PCL or collateral ligament
* Severe fixed valgus or varus deformity of >15º
* Extensor lag > 15 º
* Fixed flexion contracture ≥ 15 º
* Unwilling or unable to comply with study requirements
* Participation in another clinical study which would confound results
* Allergy to any of the implant materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
2011 Knee Society Score | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quartulli, Study Director — Restor3D; Terry Clyburn, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (9):
- United States (9):
  - JFK Medical Center, Atlantis, Florida
  - EMMC - Orthopaedic Surgery of Maine, Bangor, Maine
  - Great Lakes Bone and Joint, Battle Creek, Michigan
  - Orthopaedic Instatute of Henderson, Henderson, Nevada
  - Desert Orthopedic Center, Las Vegas, Nevada
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Advanced Orthopedics and Sports Medicine, Cypress, Texas
  - Joint Replacement Associates, Houston, Texas
  - Mansfield Orthopaedics, Morrisville, Vermont

IPD SHARING:
Plan to Share IPD: No